CLINICAL TRIAL: NCT03437889
Title: Gravity Flow Technique to Validate Proper Location of Epidural Needle Tip on Obese Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-01532
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Epidural/Anesthesia
Keywords: epidural
MeSH Terms: interventions — Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidural analgesia/anesthesia for childbirth (Experimental)
  Interventions: Other: Cold Stimulus (Ice)

INTERVENTIONS:
Other: Cold Stimulus (Ice) — The study procedure will be to use a cold stimulus (ice) to assess the subjects for hypesthesia the dermatomes of the lower abdomen between 10 and 30 minutes after the epidural catheter is inserted.

SUMMARY:
Pregnant women, with a Body Mass Index (BMI) greater than 30 kg/m2, who receive epidural analgesia/anesthesia for childbirth will have epidural catheter placement per our standard procedure, which includes using the gravity flow technique to confirm that the tip (aperture) of the epidural needle is indeed located within the epidural space. The study procedure will be to use a cold stimulus (ice) to assess the subjects for hypesthesia the dermatomes of the lower abdomen between 10 and 30 minutes after the epidural catheter is inserted. Hypesthesia to cold will be taken a sign of successful lumbar epidural block.

DETAILED DESCRIPTION:
The purpose of this study is to quantify the reliability of the gravity flow technique to accurately validate the position of the epidural needle tip when performing lumbar epidural analgesia/anesthesia for childbirth (vaginal and cesarean delivery) in women with a BMI greater than 30 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Patients requesting epidural analgesia/anesthesia for childbirth
* American Society of Anesthesiologists (ASA) physical status I to III
* Ability to speak and read English to fully comprehend the consent process
* BMI greater than 30 kg/m2

Exclusion Criteria:

* Combined spinal-epidural anesthesia
* Coagulopathy
* History of lumbar spine surgery
* Allergy or contraindication to any of the study medications
* Contraindication to epidural analgesia
* ASA physical status >III
* BMI less than 30 kg/m2

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients requesting epidural analgesia/anesthesia for childbirth
Enrollment: 100 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Measure of bilateral decrease of sensation to cold with ice | 30 Minutes Post Intervention
  Loss of sensation to ice; Following epidural procedure, subjects will be assessed to see if their epidural analgesia is working by determining if they have hyperthesia to ice on lower abdomen.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Grant, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States